CLINICAL TRIAL: NCT06440369
Title: Effets d'un Programme d'Exercice aérobie Sur cycloergomètre Chez le Patient Atteint d'Insufisance Rénale Chronique ou Polyarthrite Rhumatoïde
Brief Title: Physical Activity and Cardiovascular Risk
Acronym: PACaR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Franche-Comté (Other)
Responsible Party: Principal Investigator, Daniele Peres, Sponsor-Investigator, University of Franche-Comté
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UnivFranche-Comte
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis; Chronic Kidney Diseases; Endothelial Dysfunction; Arterial Stiffness; Exercise
MeSH Terms: conditions — Arthritis, Rheumatoid; Renal Insufficiency, Chronic; Motor Activity | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: Control group (CG): Patients will continue their lifestyle. Physical activity orientation group (G0-AP): Patients will be encouraged to practice physical activity and will benefit from telephone calls for instructions regarding this practice. They will be contacted by telephone each week, for a total of 6 calls, each lasting approximately 10 minutes.
  Training group (GE): Patients will begin the individualized PA program during the inclusion visit and will continue it for 6 weeks, at a rate of 3 sessions per week (for a total of 18 sessions). At the end, patients will be able to resume their usual activities and will be evaluated again 6 weeks after stopping the program. The training program will be supervised by a physical activity instructor adapted and carried out at the CHRU, in the Nephrology or Rheumatology Department depending on the patient's pathology.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training group (Experimental): Patients will begin the individualized physical activity program during the inclusion visit and will continue it for 6 weeks, with 3 sessions per week (for a total of 18 sessions). At the end, patients will be able to resume their usual activities and will be evaluated again 6 weeks after stopping the program. The training program will be supervised by a physical activity instructor adapted and carried out at the CHRU, in the Nephrology or Rheumatology Department depending on the patient's pathology.
  Interventions: Other: Training group
- Physical activity orientation group (Active Comparator): Patients will be encouraged to engage in physical activity and will receive phone calls for instructions regarding this practice. They will be contacted by telephone each week, for a total of 6 calls, each lasting approximately 10 minutes.
  Interventions: Other: Physical activity orientation group
- Control group (No Intervention)

INTERVENTIONS:
Other: Training group — The patient will perform an intermittent exercise which consists of nine 5-minute cycles with a succession of work (top: 1 minute; bottom: 4 minutes). The high-intensity work phase will be adjusted so as to achieve a target Heart Rate (HR) corresponding to resting HR + 80% reserve HR (reserve HR = (200 - age) - resting HR). The low-intensity work phase will be adjusted to achieve a target maximum HR corresponding to resting HR + 60% reserve HR. In total duration, the exercise presents a submaximal intensity, commonly used in exercise rehabilitation studies carried out with various pathologies. It is an intensity capable of promoting benefits on the cardiovascular aspect without representing a severe intensity for the patient.
  In order to adapt the training and guarantee patient safety, the first exercise session will be carried out with an alternation between a high-intensity work phase of resting HR + 70% reserve HR and a work phase. at low intensity of resting HR + 50% reserve HR.
  Arms: Training group
Other: Physical activity orientation group — Every week, for around ten minutes, patients in the AP orientation group will be contacted by telephone. The main objective of this exchange is to provide targeted advice on physical activity, its role, its objectives as well as its different ways of carrying it out. The second objective is to provide each week a personalized objective for each patient which can evolve over the weeks to increase levels of physical activity as far as possible. During each call, the evaluator will practice reflective listening, ask open-ended questions to facilitate the exchange, value and summarize the patient.
  Arms: Physical activity orientation group

SUMMARY:
Physical activity (PA) is essential for the prevention and treatment of chronic conditions. Despite its benefits, global physical inactivity is prevalent, contributing to chronic diseases and premature mortality. For patients with chronic kidney disease (CKD) and rheumatoid arthritis (RA), PA is particularly beneficial as it improves endothelial health, reduces cardiovascular risk, diminishes inflammation, and enhances quality of life. Given the chronic inflammation and immune system dysregulation in CKD and RA, PA may mitigate these effects and improve patient outcomes. The primary objective of this study is to evaluate the effects of a personalized aerobic exercise program on cardiovascular risk in patients with CKD or RA. The secondary objectives are to assess the effects on inflammation and immunosenescence; investigate the relationship between inflammation, immunosenescence, and various health outcomes; compare the impacts of chronic PA and PA guidance on cardiovascular risk, disease activity, lifestyle habits, cognitive functions, and quality of life.

This study presents an interventional design. A total of 105 subjects are expected to participate in this study, including 45 CKD patients and 45 RA patients. Participants will be stratified by PA level and cardiovascular risk (SCORE 2 scale) and then randomized into three groups: Control Group: 15 CKD and 15 RA patients; Therapeutic Education Group: 15 CKD and 15 RA patients; and Experimental Group: 15 CKD and 15 RA patients.

The inclusion criteria are: age > 50 years; diagnosed with CKD or RA; glomerular filtration rate between 45 and 29 ml/min/1.73 m² for CKD; DAS-28 score ≥ 2.6 for RA; medical clearance for PA; informed consent and affiliation with French social security. The exclusion criteria are: unstable corticosteroid therapy or >10 mg prednisone/day; uncontrolled hypertension; pregnancy; cognitive impairment preventing adherence to the program; inability to perform PA; legal incapacity or anticipated poor cooperation; lack of health insurance and participation in an incompatible study.

The primary efficacy criterion of this study is changes in endothelial function (macrovascular arterial stiffness) and the secondary efficacy criteria are: endothelial function (microvascular hyperemia test); levels of inflammation and immunity (blood tests); physical activity levels and quality of life (questionnaires); disease-related functional impairment; disease activity and cognitive function.

Patient screening will begin with the identification of eligible patients in the Nephrology and Rheumatology departments. Day 0 will be the selection visit for participant information and consent. A week after Day 0, the inclusion visit and initial assessment (arterial stiffness, endothelial function, disease impact, and blood markers for immunosenescence and inflammation, blood pressure, heart rate, PA level, quality of life, and cognitive functions) will be conducted for all patients. Next, only the patients in the experimental group will carry out a 47-minute cycling intermittent exercise session, perceived exertion assessment, and post-exercise reassessment. They will redo the assessments after the exercise. They will have another 16 sessions of supervised exercise by a health professional and a final session identical to the first for reassessment. Patients in the physical activity guidance group will not undertake a physical exercise program but will receive one call per week to discuss the physical activities performed and get answers to their questions on the subject. The control group will continue with their usual lifestyle habits.

DETAILED DESCRIPTION:
To address the primary objective, arterial stiffness in the experimental group will be analyzed and compared with the control group and the physical activity orientation group. To address the secondary objectives, various variables related to quality of life, cognitive functions, and disease activity will be compared between different patient groups. The levels of inflammation and immunosenescence and the relationship between these two dimensions will be analyzed before and after the exercise program in the experimental group of RA and CKD patients, with patients serving as their own controls.

The first contact with CKD patients will be in the Nephrology Department, and for RA patients, in the Rheumatology Department during their regular medical visits. Initially, investigators will screen potential patients for participation. The screening process involves a thorough evaluation of medical characteristics, health history, and other pre-established criteria to identify subjects who meet the specific inclusion criteria of this study.

The evaluations described in the initial assessment will be conducted, and all enrolled subjects will undergo a resting ECG, with the investigator recording data for each subject. Patient treatments will not be interrupted during the entire protocol period. All patients will be evaluated twice: once during the inclusion visit and again after 6 weeks.

During the inclusion visit, the patient will complete questionnaires, then rest in a lying position for 10 minutes. An initial evaluation lasting about 10 minutes will be conducted in a lying position, including measurements of blood pressure, heart rate, reactive hyperemia (to evaluate endothelial function), and pulse wave velocity (PWV). The total duration will be 25 minutes. After then, for control group patients and physical activity orientation group patients, the session ends here.

For experimental group patients, the patient will then perform physical activity on a cycle ergometer for 47 minutes. The same assessments will be conducted at the end of the session For invasive measures, venous blood samples will be taken from the elbow crease by a clinical research nurse. A total of 2 dry tubes of 5 ml and 2 EDTA purple tubes of 5 ml will be collected at the beginning and end of the rehabilitation protocol (6 weeks), totaling 40 ml. For experimental groups, an additional blood sample will be taken during follow-up, 6 weeks after the end of the rehabilitation program, totaling 60 ml for these groups.

Endothelial function will be assessed by measuring pulse wave velocity and reactive hyperemia. Arterial compliance (central and peripheral) will be assessed by measuring the pulse wave velocity on the carotid-femoral and carotid-radial segments, respectively, using the Complior (Complior SP®, Artech Medical, Pantin, France). Reactive hyperemia will be assessed with ENDOPAT (Itamar Medical®, Caesarea, Israel), which quantifies peripheral vasodilatory response non-invasively via electronic finger cuffs following blood flow occlusion.

Hemodynamic parameters will be evaluated by measuring heart rate and blood pressure with the Finapres during assessments. Heart rate monitoring during cycling in experimental groups will use the Polar A300 heart rate monitor. Blood pressure will be measured before and after exercise with the Omron.

The interventions during the 6 weeks for the experimental group - exercise sessions will be conducted in the nephrology or rheumatology departments, supervised by an adapted physical activity professional, scheduled for three weekly 47-minute sessions over 6 weeks (18 sessions). Exercise intensity will be adjusted based on individual heart rate reserve, starting at 40% and progressing to 70% by the final session. Each session includes a warm-up, main exercise phase, and active recovery.

The interventions during the 6 weeks for the PA orientation group - Every week, for around ten minutes, patients in the PA orientation group will be contacted by telephone. The main objective of this exchange is to provide targeted advice on physical activity, its role, its objectives as well as its different ways of carrying it out. The second objective is to provide each week a personalized objective for each patient which can evolve over the weeks in order to increase levels of physical activity as far as possible. Call Procedure are: establishing a diagnosis carried out using questionnaires distributed beforehand (level of physical activity, quality of life); contribution of advice and explanation around physical activity: The evaluator (adapted physical activity teacher) will provide knowledge about PA, its roles and objectives, recommendations, and different ways of practice; lifestyle exchange (personalized): An exchange between the professional and the patient to understand the patient's lifestyle habits; setting a therapeutic objective: Propose an objective around physical activity based on the patient's needs and lifestyle and answer patient questions: Reflective listening and open-ended questions will facilitate the exchange.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject (man or woman) over 50 years old, without diagnosis of chronic disease.
* Patient (man or woman) over 50 years old, with a diagnosis of CKD or RA without other risk factors related to the disease.
* Have a medical certificate of no contraindication to AP.
* Have a glomerular filtration rate between 45 and 29 ml/min/1.73 m2, corresponding to non-dyalized stages III and IV for patients with CKD.
* Have a DAS-28 score ≥ 2.6 points for patients with RA.
* Signature of informed consent.
* Affiliation to a French social security scheme or beneficiary of such a scheme.

Exclusion Criteria:

* unstabilized corticosteroid therapy and/or >10 mg of prednisone/day;
* unbalanced high blood pressure;
* pregnant women ;
* alteration of higher functions making understanding and adherence to a conditioning program impossible;
* inability to perform physical exercise, whatever the origin (neurological, central or peripheral, cardiac, vascular or respiratory or musculoskeletal).
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject without health insurance
* Subject being in the period of exclusion from another study or provided for by the "national volunteer file".

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  The evaluation of central and peripheral arterial compliance will be carried out by measuring the pulse wave velocity on the carotid-femoral and carotid-radial segments respectively. These evaluations are carried out using the Complior device (Complior SP®, Artech Medical, Pantin, France). This system is equipped with an interface between the piezoelectric sensors and the laptop which is used to save the recordings. The search for the best site at the radial, femoral and carotid levels will be done by palpation. Once the sites have been identified, the operator will mark them using a hypoallergenic marker so as to find the same measurement positions during the session (for the experimental and healthy group). The sensors will be held in place with a velcro system or by the operator. After checking the quality of the signal and after leaving the subject to rest for a few minutes, the operator can record the signal.
Reactive hyperemia | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  The evaluation of the hyperemic reaction will be carried out by ENDOPAT (Itamar Medical®, Caesarea, Israel). This tool quantifies the peripheral vasodilator response (reactive hyperemia) via an electronic finger cot in a non-invasive manner, following occlusion of vascular flow. The measuring device is made up of two probes with an inflation system placed on the index finger of each hand. On the side of the finger tested, after measuring the basal flow, a cuff positioned at the level of the arm is inflated above the systolic pressure for 5 minutes, then released creating a reflex vasodilation measured by the ENDOPAT. Endothelial function is calculated by the relationship between the average amplitude of reactive hyperemia over a 1 minute period starting 1.5 minutes after cuff deflation and the baseline level.

SECONDARY OUTCOMES:
Inflammation level | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  Venous blood samples will be used to measure CD4 and CD8 concentrations and IL6 concentrations; CRP; TNF-α.
Level of quality of life | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  The Short Form 36 (SF-36) health survey questionnaire is the most commonly used generic instrument to assess health-related quality of life in the general population. This questionnaire validated in French was developed by Ware and Sherbourne in 1992 based on the Medical Outcome Study. The questionnaire consists of 36 questions assessing the following 8 dimensions: physical activity, physical limitations, physical pain, perceived state of health, life and relationships with others, limitations due to physical state , mental health and finally a comparison with the state of health perceived one year previously. This questionnaire was selected because of its speed of administration (around ten minutes), its self-administrability and its ease of use. The range is 0 to 100 points, where higher scores indicate better physical functioning.
Level of physical activity | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  The PA level will be measured by the short version of the "International Physical Activity Questionnaire - IPAQ". This questionnaire makes it possible to assess overall physical activity and the level of sedentary lifestyle during the last seven days of patients. The IPAQ questionnaire therefore focuses on the practice of intense, moderate activities, walking, and the time spent sitting (sedentary lifestyle), whether during leisure activities, at work, in daily life or again during transport. The short version of the IPAQ questionnaire validated in French includes 7 questions. The questionnaire thus makes it possible to classify the subject according to 3 activity levels: inactive, moderate and high. This questionnaire was selected because of its speed of administration (less than 10 minutes) and its ease of use. The range varies depending on the person's activities, with higher scores indicating higher levels of physical activity.
Systolic pressure (mmHg) and diastolic pressure (mmHg) | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  They will be measured continuously at the finger using the photoplethysmographic method on the non-dominant side (Finapres, Finapres Medical Systems, Amsterdam). The Finapres method is a non-invasive technique that measures beat-to-beat variations in blood pressure and heart rate. It was validated against intra-arterial recordings as well as the traditional blood pressure monitor
Heart rate (HR, bpm) | Assessment on the same day of the inclusion visit and 6 consecutive weeks later.
  They will be measured continuously at the finger using the photoplethysmographic method on the non-dominant side (Finapres, Finapres Medical Systems, Amsterdam). The Finapres method is a non-invasive technique that measures beat-to-beat variations in blood pressure and heart rate. It was validated against intra-arterial recordings as well as the traditional blood pressure monitor

IPD SHARING:
Plan to Share IPD: Undecided